CLINICAL TRIAL: NCT06271213
Title: The Gut-Lung Axis and Respiratory Illness in Children
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: 303841
Record Dates: First submitted 2024-01-30; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Respiration Disorders; Respiratory Disease; Asthma in Children; Wheezing; Gastro-Intestinal Disorder; Healthy
Keywords: Gut-Lung Axis; Microbiome; Multi-omics; Children
MeSH Terms: conditions — Respiration Disorders; Respiratory Sounds; Digestive System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Nasopharyngeal swabs immunological/metabolic/microbiome analyses Lower airway Samples for immunological/metabolic/microbiome analyses stool samples for immunological/metabolic/microbiome analyses blood samples for for immunological/metabolic analyses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Respiratory Disease: Children with respiratory complications receiving general anaesthesia undergoing bronchoscopy
  Interventions: Other: observational only - no interventions as part of study
- Gastrointestinal Disease: Children with G.I. complications receiving general anaesthesia undergoing endoscopy
  Interventions: Other: observational only - no interventions as part of study
- Orthopaedic controls: Children with orthopaedic issue receiving general anaesthesia undergoing orthopaedic correction
  Interventions: Other: observational only - no interventions as part of study
- Asthma Control: Children with Asthma/wheeze not indicated for biologics therapy
  Interventions: Other: observational only - no interventions as part of study
- Asthma Treatment: Children with Asthma/wheeze indicated for biologics therapy
  Interventions: Other: observational only - no interventions as part of study

INTERVENTIONS:
Other: observational only - no interventions as part of study — Children with asthma will be receiving biologics therapy as part of their standard of care - unrelated to this study design. All cohorts will be observed without study intervention.

SUMMARY:
The goal of this single-centre observational study conducted at the Royal Hospital for Children in Glasgow, Scotland, is to employ a multi-omics approach to investigate the "gut-lung axis" in health and disease.

Part A is a cross-sectional study design investigating the postulated bidirectional link between the gut and lung microbiomes in children suffering from respiratory or gastrointestinal conditions. Children with no GI or respiratory issues attending for orthopaedic care will be used as a benchmark for a healthy gut-lung axis. The main questions we aim to answer are:

* What does a healthy gut-lung axis look like?
* Do children with respiratory issues show an altered gut microbiome?
* Do children with GI issues show an altered lung microbiome?

Part B is a longitudinal study design, that aims to assess the effects of biologics on the gut-lung axis by comparing the gut and lung microbiomes in children with asthma at two time-points who are indicated to start biologics therapy (Asthma treatment) or will not receive biologics therapy (asthma control).

Participants will provide:

* airway samples (to investigate the lung microbiome)
* blood samples (to assess inflammatory and metabolic factors which may mediate communication between the two sites) whilst under general anaesthetic for a treatment related to their standard of care
* stool samples (to assess gut microbiome)
* dietary information (food diary and/or food frequency questionnaire) to assess relationships between diet and the gut-lung axis.

DETAILED DESCRIPTION:
The gut-lung axis is a postulated bi-directional connection between the gut and lung microbiomes where changes at one site can induce changes in another. Although pre-clinical evidence exists, the clinical evidence, particularly in paediatric patients is currently lacking. Changes in the gut microbiome in young children have been noted prior to asthma development although concomitant investigations into the gut and lungs have not yet been made in children with asthma. Furthermore, a causal relationship between IBD and respiratory disease has recently been noted. Associations have also been made between early-life environmental factors such as the protective effects of breastfeeding on respiratory health which hints at connections between dietary intake and respiratory health, possibly via the gut-lung axis. The investigators aim to investigate the gut-lung axis in children via a multi-omics approach.

Part A (cross-sectional): The investigators aim to investigate correlations between the gut and lung microbiome in 3 cohorts of children aged 0-16 attending the Royal Hospital for Children in Glasgow: Respiratory patients, GI patients and Orthopaedic patients. Although this is a hypothesis-generating study, the investigators would like to validate this bi-directional link between the gut and the lung microbiomes. The investigators hypothesise that children with respiratory disease should have a disturbed gut microbiome and children with GI disease should present with a disturbed respiratory microbiome (assessed ecologically and functionally via metabolic and molecular biology analyses). Children receiving orthopaedic procedures without active signs of respiratory or GI issues will serve as the benchmark of a healthy 'gut-lung axis'. The investigators will also aim to investigate potential mechanisms of communication between the gut and lungs in blood via immunological, metabolic, and molecular analyses. Dietary analysis, relevant clinical data and a health questionnaire will be completed by children. Additionally, a 3-day estimated weighed food diary will be completed by the participants and a validated Food Frequency Questionnaire (FFQ) in children aged 3 and above will be used to correlate dietary intake to biological date obtained relating to the gut-lung axis.

Part B (longitudinal): Investigating the Gut-Lung axis in asthma pre and post biologics therapy. The investigators aim to investigate connections between the airway and gut-microbiome, blood and responsiveness to patients receiving biologics therapy (as part of their standard of care). Two cohorts of children will be recruited: children with asthma/wheeze not indicated for biologics and children with asthma/wheeze indicated for biologics. The investigators aim to assess whether biologics modulate the gut-lung axis by sampling airways, stool and blood from children at two time points (before and after starting therapy, compared to the no therapy group). Nutritional data and relevant clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Any infant/child/young person admitted to the RHC, Glasgow for an elective bronchoscopy or GI endoscopy.
* Any infant/child attending for an emergency/elective orthopaedic operation without active respiratory or gastrointestinal conditions or receiving treatment for either condition. (Age range birth to 16 years for all groups recruited).
* Any child attending respiratory department at RHC who can induce sputum and is having a blood sample taken, with latter part of standard of care.
* Any infant/child/young person admitted to RHC for a clinical care appointment with Asthma/wheeze before commencement of biologics therapy (treatment group).
* Any child admitted to RHC with asthma/wheeze not indicated for biologic therapy (asthma control group).

Exclusion Criteria:

* Use of antibiotics by the day of admission or have used antibiotics in the previous month (unless prophylactic antibiotics > 1 month use).
* Any person 17 years old and above.
* Any child known to be infected with, or at high risk of having had exposure to HIV, hepatitis B or hepatitis C viruses
* . Any child and/or parent/guardian who cannot understand the English language where consent would be unethical.
* Any child with Asthma currently receiving Biologics therapy (unless recruited via bronchoscopy route).

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children attending Royal Hospital for Children, Glasgow receiving general anaesthesia for bronchoscopy, endoscopy or orthopaedic procedures. Children attending Royal Hospital for Children for routine procedures with asthma/wheeze.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Assess differences in gut and lung microbiota diversity between groups | At admission on a single day
  Beta diversity: measure the differences in species composition between different ecosystems. Are there statistically significant differences in beta-diversity (p<0.05 between the gut and airway microbiome of cohorts)
Assess changes in gut and lung microbiota in children with asthma receiving biologics | Measurement 1 at baseline. Measurement 2 anywhere from 8-52 weeks.
  Alpha diversity: measure of species richness and evenness within a sample. Are there statistically significant (p<0.05) differences in species richness and evenness at sampled anatomical sites between cohorts.
Determine mediators of gut-lung axis in health and disease | At admission on a single day. Between Timepoints A (baseline) and B (from 8-52 weeks) in asthma arm.
  Are there statistically significant differences (p<0.05) in immunological/nutritional/metabolic/transcriptional factors in health and disease

SECONDARY OUTCOMES:
Nutritional influence in gut-lung axis | approximately up to 12 weeks before to 12-weeks after admission.
  Correlations between dietary factors (assessed via dietary questionnaires and/or food diary) on the gut-lung axis.
Multi-omics integration | At admission on a single day. Between Timepoints A (baseline) and B (from 8-52 weeks) in asthma arm.
  Can a multi-omics view enhance our understanding of the gut-lung axis by integrating microbiome, immunological and nutritional/metabolic data.

CONTACTS AND LOCATIONS:
Overall Officials: Ross J Langley, MRCPCH, Principal Investigator — NHS Greater Glasgow and Clyde Board HQ
Locations (1):
- NHS Greater Glasgow and Clyde: Royal Hospital for children, Glasgow, Glasgow, United Kingdom